CLINICAL TRIAL: NCT02451345
Title: Development, Validation, and Dissemination of an Integrated Risk Prediction Model and Decision Aid to Discern Aggressive vs Indolent Prostate Cancer (Aim 2A)
Brief Title: Decision Support Tools for Men With Prostate Cancer- Clinical & Lifestyle Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14557; NCI-2018-02056 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Tranformative Impact Award; Early stage; Active Surveillance; Decision aid; Coaching session; Personalized; UCSF; validation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Personalized risk model+website+phone coaching
  Interventions: Behavioral: Personalized risk model+website+coaching intervention

INTERVENTIONS:
Behavioral: Personalized risk model+website+coaching intervention — A health coach (members of the Patient Support Corps at the University of California San Francisco) will contact each subject individually to discuss his tailored/personalized web-portal report on his risk of aggressive disease and the pro/cons of treatment versus active surveillance.
  The contact between subject and the health coaches will be done before subject's visit with his primary urologist. Subjects will be asked to complete different questionnaires on four different occasions: one at first visit to the interactive secure web portal; one before coach's call; one after the coaching (after the urologist visit), and one at 6 months. The questionnaire after subject's visit with the urologist includes discussion about their management choice, decision quality, anxiety and satisfaction with care.

SUMMARY:
A UCSF PI-initiated study with a primary goal to improve decision quality, anxiety, and uncertainty, thereby increasing appropriate uptake of active surveillance and reducing over-treatment of low-risk prostate cancer.

This study involves: completion of questionnaires through the secure website; consultation by a health coach to aid men with prostate cancer in making informed treatment decision (personalized coaching session(s)).

DETAILED DESCRIPTION:
A UCSF PI-initiated study which includes comprehensive decision support intervention that may incorporate clinical, lifestyle, tumor genomic, and germline gene variant data.

The web and coaching intervention will: 1) summarize key prognostic data elements, 2) communicate relative and absolute risks of upgrading/upstaging based on each of these elements, individually and in aggregate, and 3) provide tailored educational information for informed decision making on treatment options. A key aspect of the intervention will be provision of tiered coaching to the men prior to their physician visits to help them enter information accurately into the system, understand the results of the prediction model, document their questions for their physicians, and prepare them to make better-informed treatment decisions. UCSF research team will develop the decision support intervention in phases, initially using only clinical variables, BMI (body mass index), and smoking data;and then extend it to include information from genomic and genetic inputs, as validation work progresses. Variables will be retained based on statistical evaluation of the predictive values.

ELIGIBILITY:
Inclusion criteria are the following:

1. Men >18 years of age with newly diagnosed (within 3 month) low risk prostatecancer , who have not yet received cancer-directed therapy, Or Men who are at risk of prostate cancer and coming to have a diagnostic biopsy, and diagnosed with low grade of prostate cancer
2. Biopsy Gleason score < 3+3,
3. Has localized (clinical stage < T2N0M0) prostate cancer with a PSA <10ng/ml
4. Consent to research follow-up

Exclusion Criteria:

1. men with missing data on PSA, stage, Gleason, or extent of biopsy core involvement; no baseline (diagnostic) biopsy or germline DNA sample for research; or no follow-up pathology (from biopsy or RP) after diagnosis.
2. men unable to consent, prisoners, those with ECOG performance status >2, or psychiatric illness/social situations that would limit compliance with study requirements, or inability to read English or Spanish.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Decision Quality measured using the Decision Quality Index | 12 months
  measured using the Decision Quality Index

SECONDARY OUTCOMES:
Prostate Cancer Specific Anxiety measured using MAXPC survey | 12 months
  Measured using MAXPC survey
Decision Self- Efficacy measured using Decision Self-Efficacy survey | 12 months
  Measured using Decision Self-Efficacy survey

CONTACTS AND LOCATIONS:
Overall Officials: Peter Carroll, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of California, San Francisco (SFGH), San Francisco, California

IPD SHARING:
Plan to Share IPD: No